CLINICAL TRIAL: NCT01920399
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety, Tolerability and Pharmacokinetics of Ceftazidime-Avibactam Administered as Single and Repeated Intravenous Doses in Healthy Chinese Subjects
Brief Title: A Phase I Study to Assess the Safety, Tolerability and PK of Ceftazidime-Avibactam in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: D4280C00020
Record Dates: First submitted 2013-07-25; First posted 2013-08-12 (Estimated); Last update posted 2017-09-05 (Actual); Status verified 2017-09

CONDITIONS: Healthy Volunteers
Keywords: CAZ-AVI China phase I PK study
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): IV infusions of 0.9% normal saline
  Interventions: Drug: 0.9% Normal Saline
- CAZ-AVI (Experimental): IV infusion of AVI 500 mg + CAZ 2000 mg.
  Interventions: Drug: CAZ-AVI

INTERVENTIONS:
Drug: CAZ-AVI — A single 120 minute IV infusion on Day 1, followed by three times daily (every 8 hours, q8h) as 120 minute IV infusions for 7 days (Day 2 to Day 8), and one single 120 minute IV infusion on Day 9.
  Arms: CAZ-AVI
Drug: 0.9% Normal Saline — A single 120 minute IV infusion on Day 1, followed by three times daily (every 8 hours, q8h) as 120 minute IV infusions for 7 days (Day 2 to Day 8), and one single 120 minute IV infusion on Day 9.
  Arms: Placebo

SUMMARY:
Investigate the safety and tolerability, as well as PK profile of ceftazidime-avibactam (CAZ -AVI) administered in single and repeated intravenous (IV) infusions in healthy Chinese subjects.This study data will be used to support CAZ-AVI NDA in China.

ELIGIBILITY:
Key Inclusion Criteria:

* Provision of signed and dated, written informed consent prior to any study-specific procedures.
* Healthy male and female (of non-child bearing potential) Chinese subjects, with suitable veins for cannulation or repeated venipuncture
* BMI 19 to 24 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg.

Key Exclusion Criteria:

* Any clinical condition requiring the regular use of any medication.
* Consumption of alcohol, drug, tobacco (cigarettes).
* Sensitive to any food, or any serious reaction to carbapenem, cephalosporin, or other β-lactam antibiotics.
* Severe medical or psychiatric condition or laboratory abnormality.
* Blood donation.
* 12 lead ECG abnormal.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2013-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability:Adverse events, vital signs, ECGs, clinical laboratory measurements, physical examinations, oral body temperature | Routine safety assessments, throughout the period that subjects receive CAZ-AVI/PLACEBO up to 5 days following discontinuation of study treatment
  AE: The onset of an AE relative to treatment will be calculated as the time difference between the onset (date and time) of the AE and the start time of the last dose (date and time) prior to the AE; the duration of a resolved AE will be calculated as the difference between the resolution (date and time) of the AE and the onset (date and time) of the AE. Vital signs and oral temperature:Change in BP, pulse rate and oral temperature at each post treatment time point will be calculated as the post treatment measurement value minus the baseline value observed on Day -1. Physical examination: complete physical examination and brief physical examination. ECG: heart rate, RR, PR, QRS, and QT intervals from the 12-lead ECG and the derived variable QTcF. Safety laboratory (hematology, chemistry and urinalysis): Change in laboratory test value at each post treatment time point will be calculated as the post treatment value minus the baseline value observed on Day -1 .

SECONDARY OUTCOMES:
Plasma PK parameters for CAZ and AVI of single dose: Cmax, tmax, Clast, tlast, AUC(0-t), AUC, AUC(0-8), λz, t1/2, Vss, Vz, CL, MRT, etc. | single IV infusion on Day 1
Plasma PK parameters for CAZ and AVI of multi dose: the trough concentration Cmin | Days 6, 7, 8
Plasma PK parameters for CAZ and AVI of repeated infusion: Cmax, tmax, Clast, tlast, AUC(0-t), AUC, AUC(0-8), λz, t1/2, Vss, Vz, CL, MRT, etc. | After repeated infusion On Day 9
Urine PK parameters for CAZ and AVI of single and repeated infusion: Cumulated urinary excretion (amount), percentage of cumulated urinary recovery (% dose) and renal clearance (CLr) | Day 1 and Day 9

CONTACTS AND LOCATIONS:
Overall Officials: Furong Qiu, Principal Investigator — Shuguang Hospital affiliated with Shanghai University of TCM
Locations (1):
- Research Site, Shanghai, China

REFERENCES:
- [Background] Li J, Learoyd M, Qiu F, Zhu L, Edeki T. A Randomized, Phase I Study to Assess the Safety, Tolerability and Pharmacokinetics of Ceftazidime-Avibactam in Healthy Chinese Subjects. Clin Drug Investig. 2016 Feb;36(2):119-26. doi: 10.1007/s40261-015-0347-x. PMID 26649741
- [Derived] Li J, Lovern M, Green ML, Chiu J, Zhou D, Comisar C, Xiong Y, Hing J, MacPherson M, Wright JG, Riccobene T, Carrothers TJ, Das S. Ceftazidime-Avibactam Population Pharmacokinetic Modeling and Pharmacodynamic Target Attainment Across Adult Indications and Patient Subgroups. Clin Transl Sci. 2019 Mar;12(2):151-163. doi: 10.1111/cts.12585. Epub 2018 Sep 28. PMID 30221827
- See also: D4280C00020_Revised_CSP_1_redacted_protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1834&filename=D4280C00020_Revised_CSP_1_redacted_protocol.pdf